CLINICAL TRIAL: NCT03545724
Title: Prospective, Single Arm, Open Study to Evaluate the Effect of NeoFitoroid® in Reducing Symptoms in Patients With Hemorrhoidal Disease
Brief Title: Effectiveness & Safety of Neofitoroid® in Hemorrhoidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: GB Pharma Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABO-NFT-17
Record Dates: First submitted 2018-05-21; First posted 2018-06-04 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2018-05

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neofitoroid® (Experimental): Treatment is made by the application of Neofitoroid® 2 times a day for 10 days.
  Interventions: Device: Neofitoroid®

INTERVENTIONS:
Device: Neofitoroid® — NeoFitoroid® forms a protective barrier mucosa and on perianal region that can aid the physiological process of healing.
  Other Names: Rescue therapy

SUMMARY:
Evaluation of the effect and safety of NeoFitoroid® in reducing symptoms in patients with hemorrhoidal disease.

DETAILED DESCRIPTION:
Evaluation of the effect and safety of NeoFitoroid® in relieving discomfort symptom after 10 days of treatment compared to baseline (pretreatment).

The study duration per patient is 31 days (visit 1 + 10 days treatment + 20 days follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes ≥ 18 years .
2. Diagnosis of hemorrhoidal disease of grade I or II, non thrombosed, according to Goligher's classification performed by anoscopy/rectoscopy at screening.
3. Patient is not expected to require non-pharmacological (as Sclerotherapy, Rubber band ligation, Infrared Coagulation, Radiofrequency Ablation, Cryotherapy) or surgical treatment in the 31 days post enrollment .
4. Discomfort score related to the hemorrhoidal disease ≥ 30 measured through a 0-100 Visual Analog Scale VAS (from "no symptoms" to "overwhelming symptoms") at screening.
5. Women of childbearing potential undergone a negative pregnancy test.
6. Informed consent documentation signed and dated confirming that the patient has been adequately informed of all aspects related to his/her participation in the clinical study and is willing to participate.

Exclusion Criteria:

1. Patients with gastrointestinal disease like inflammatory bowel disease, celiac disease, colo-rectal cancer, perianal/fistulizing disease).
2. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and/or that, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
3. Patients with active cancer.
4. Tubercolosis , mycosis, Herpes Symplex, virologic disease with anal or perianal skin localization.
5. Presence of physical and/or mental disability that reduces the ability to take medicines as expected.
6. Concomitant abuse of drugs or alcohol.
7. No adequate reliability or presence of conditions that may result in non-compliance / adherence of the patient to the Protocol.
8. Subjects with known or suspected allergy to plants of Helichrysum family, aloe vera, Ruscus, Hypericum, Jojoba Oil, Shea Butter, Essential oils of: Melaleuca, Cypress and Peppermint.
9. Subjects with known or suspected allergy to ingredients such as: glicerilstearato, Caprylic / capric, sucrose distearate, sucrose stearate, cetearyl alcohol, vegetable glycerin, triidrossistearina, vegetable oils, hydrogenated vegetable oils, Candelilla wax, xanthan gum, citric acid, tocopherols, sodium silicate, benzyl alcohol, potassium sorbate, sodium dehydroacetate, Sunflower oil.
10. Subjects with the presence of alarm symptoms (weight loss, lack of appetite).
11. Prior use of other topical ointment for the treatment of haemorrhoid within 14 days before enrollment.
12. Pregnant and/or breastfeeding patients.
13. Participation in interventional research studies of investigational medicinal or device products (ongoing or terminated less than 30 days before screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Neofitoroid® in relieving discomfort symptoms after 10 days of treatment compared to baseline (pretreatment). | day 10 vs day 0
  Reduction of discomfort symptoms measured through a 0-100 Visual Analog Scale related to hemorrhoidal discomfort (VAS, from "no symptoms" to "overwhelming symptoms", 100-mm scale) after 10 days of treatment compared to baseline.
  The higher values represent a worse outcome. Primary endpoint will be evaluated only with the hemorrhoidal discomfort VAS

SECONDARY OUTCOMES:
Relief in discomfort symptom at 3 and 7 days of treatment compared to baseline (pretreatment). | day 3 and day 7 vs day 0
  To evaluate the Reduction of discomfort symptom measured through a 0-100 Visual Analog Scale related to hemorrhoidal discomfort (VAS, from "no symptoms" to "overwhelming symptoms", 100-mm scale). The higher values represent a worse outcome. This secondary endpoint will be evaluated only with the hemorrhoidal discomfort VAS
Relief in pain symptom at 3, 7 and 10 days of treatment compared to baseline (pretreatment). | day 3, day 7 and day 10 vs day 0
  To evaluate the Reduction of pain symptom measured through a 0-100 Visual Analog Scale related to hemorrhoidal pain symptom (VAS, from "no symptoms" to "overwhelming symptoms", 100-mm scale). The higher values represent a worse outcome. This secondary endpoint will be evaluated only with the hemorrhoidal pain symptom VAS
Relief in itching at 3, 7 and 10 days of treatment compared to baseline (pretreatment). | day 3, day 7 and day 10 vs day 0
  Reduction of itching symptoms measured through a 0-100 Visual Analog Scale related to hemorrhoidal itching (VAS, from "no symptoms" to "overwhelming symptoms",100-mm scale). The higher values represent a worse outcome. This secondary endpoint will be evaluated only with the hemorrhoidal itching VAS
Relief in burning at 3, 7 and 10 days of treatment compared to baseline (pretreatment). | day 3, day 7 and day 10 vs day 0
  Reduction of burning symptoms measured through a 0-100 Visual Analog Scale related to hemorrhoidal burning (VAS, from "no symptoms" to "overwhelming symptoms", 100-mm scale). The higher values represent a worse outcome. This secondary endpoint will be evaluated only with the hemorrhoidal burning VAS
Absolute reduction of discomfort pre and post defecation at 3, 7, and 10 days of treatment compared to baseline (pretreatment). | day 3, day 7 and day 10 vs day 0
  Absolute reduction of discomfort pre and post defecation measured through a 0-100 Visual Analog Scale related to hemorrhoidal discomfort (VAS, from "no symptoms" to "overwhelming symptoms", 100-mm scale). The higher values represent a worse outcome. This secondary endpoint will be evaluated through a compiled VAS pre-defecation and a compiled VAS post-defecation. This secondary endpoint will be evaluated through mean of the differences (VAS score post-defecation - VAS score pre-defecation) at differents time of study compared to the mean measured at baseline.
Reduction of bleeding at 3, 7 and 10 days of treatment compared to baseline (pretreatment). | day 3, day 7 and day 10 vs day 0
  To evaluate the Reduction of bleeding as measured by a 6 point scale (never, rarely, sometimes, often, very often, always) for bleeding.
Reduction of anal leakage at 3, 7 and 10 days of treatment compared to baseline (pretreatment). | day 3, day 7 and day 10 vs day 0
  To evaluate the Reduction of anal leakage measured by a 6 point scale (never, rarely, sometimes, often, very often, always) for bleeding
Evaluation of presence of prolapse and/or nodules after 10 days of treatment compared to baseline (if present) | day 10 vs day 0
  To evaluate the Presence of prolapse and/or nodules after 10 days of treatment
Subject quality of life (EQ-5D-5L improvement after 10 days of treatment compared to baseline (pretreatment). | day 10 vs day 0
  To evaluate the Quality of life improvement measured with Quality of Life Index (EQ-5D-5L, MOVEMENT CAPACITY, PERSONAL CARE, LIVING ACTIVITIES, PAIN OR DISCOMFORT, ANXIETY OR DEPRESSION). The higher values represent a worse outcome.

OTHER OUTCOMES:
Assessment on number of defecation at day 0, 3, 7 and 10. | day 3, day 7 and day 10 vs day 0
  To evaluate the Assessment on number of defecation
Assessment on type of defecation at day 0, 3, 7 and 10. | day 3, day 7 and day 10 vs day 0
  To evaluate the Assessment on type of defecation (normal, constipated or diarrheal)
Assessment of number of relapses between end of treatment and day 31 | day 31 vs day 10
  To evaluate the Number of relapses assessed between end of treatment and day 31, through patient telephone interview.
Safety and tolerability: analysis of adverse events and serious adverse events | from day -7 to day 31
  To evaluate safety and tolerability of NeoFitoroid® through the analysis of adverse events and serious adverse events that will be recorded throughout the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Patologie del Tratto Alimentare, S. Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No